CLINICAL TRIAL: NCT00819793
Title: Thoratec CentriMag VAS Failure-to-Wean From Cardiopulmonary Bypass Trial
Brief Title: CentriMag Ventricular Assist System in Treating Failure-to-Wean From Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXP-002
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: Cardiac Dysfunction; Failure-to-wean from CPB; CentriMag; Levitronix; Thoratec Corporation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CentriMag Ventricular Assist System (Experimental): All patients meeting the patient selection criteria will be treated with the CentriMag Ventricular Assist System.
  Interventions: Device: CentriMag Ventricular Assist System

INTERVENTIONS:
Device: CentriMag Ventricular Assist System — All eligible subjects will receive the CentriMag Ventricular Assist System. The system is comprised of a single-use centrifugal blood pump, a motor, a primary drive console, a back up drive console and cannulae. Blood from the failing heart is directed from the ventricle or the atrium to the inlet of the pump via an inlet cannula. Blood exits through the outlet port of the pump through the outlet cannula ultimately to the pulmonary or systemic circulation. The system can be used in either a right, left or biventricular configuration.

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the CentriMag ventricular assist system to help patients who have experienced heart failure during surgery and cannot be removed from cardiac bypass.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Cardiac dysfunction due to failure-to-wean from cardiopulmonary bypass
* Subjects who are on IABP, CPB, ECMO or CPS support prior to evaluation should have the device turned off, if possible, for the purpose of measuring inclusion hemodynamics. However, these devices should not be turned off in patients who would be harmed by interruption of support.
* All subjects must meet the following criteria at the time of enrollment:
* Hemodynamics:

  1. cardiac index ≤ 2.2 L/min/m2
  2. For patients being evaluated for left-sided support (LVAD): PCWP ≥ 18 mmHg or PADP ≥ 18 mmHg or LAP ≥ 18 mmHg
  3. For patients being evaluated for right or biventricular support: CVP ≥ 15 mmHg or RAP ≥ 15 mmHg and RVSWI ≤ 4.1 gm/m2/beat
  4. Enrollment without hemodynamic measurements due to frequent or unpredictable dysrhythmias, unacceptable cardiac function, or hemodynamic instability is allowed.
* Placement of an intra-aortic balloon pump has been attempted unless contraindicated
* All possible measures have been attempted to correct low arterial pH, arterial blood gas abnormalities, electrolytes, hypovolemia, hypervolemia, inadequate cardiac rate, dysrhythmias and residual hypothermia
* Cardiac resuscitation using pharmacologic agents, and epicardial pacing (if appropriate and possible) has been attempted
* Written, signed, and dated informed consent

Exclusion Criteria:

* BUN > 100 mg/dl
* Creatinine > 5 mg/dl
* Presence of any investigational mechanical circulatory support device
* Known history of liver cirrhosis or portal hypertension
* Pulmonary infarction
* Stroke, TIA or history of either condition within the last six months and/or any confirmed, existing neurologic deficits
* Active systemic infection defined as positive blood cultures, core temperature >100.5 degrees, white blood count > 12,500, and treatment with antimicrobials
* Participation in a clinical trial with any experimental treatment within 30 days prior to screening or previous participation in the present study
* Other serious disease(s) limiting life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Abbott Medical Devices
Locations (14):
- United States (14):
  - Mayo Clinic Hospital, Arizona, Phoenix, Arizona
  - Yale University, New Haven, Connecticut
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Fairview University Medical Center, Minneapolis, Minnesota
  - New York Columbia Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - St. Luke's Episcopal, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol included an enrollment allowance of 30 subjects at 25 centers for subjects who fail to wean from cardiopulmonary bypass. 2 additional patients were enrolled to increase the number of LVAD use in the study. Subject enrollment commenced in October 2008. A total of 18 sites participated in the study.
Groups:
- Patients Supported by the CentriMag Ventricular Assist System: All patients meeting the patient selection criteria will be treated with the CentriMag Ventricular Assist System.
  Blood from the failing heart is directed from the ventricle or the atrium to the inlet of the pump via an inlet cannula. Blood exits through the outlet port of the pump through the outlet cannula ultimately to the pulmonary or systemic circulation. The system can be used in either a right, left or biventricular configuration.
Period: Overall Study
Arm/Group | Patients Supported by the CentriMag Ventricular Assist System
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CentriMag Ventricular Assist System
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 24
Medical History [Count of Participants; unit: Participants] — Prior Cardiovascular Events examples include Arrhythmias, Valve repair or replacement, myocardial infarction, coronary artery bypass grafting (CABG), etc.
  Participants
    Smoking | 14
    Diabetes | 12
    Hyperlipidemia | 16
    Prior Cardiovascular Events | 29
Ethnicity/Race [Count of Participants; unit: Participants]
  African American | 4
  Asian | 0
  Hispanic | 2
  Native American | 0
  White | 24
  Other | 2
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 91.1 (21.4)
Laboratory Values [Mean (Standard Deviation); unit: mg/dl] — Population: Some lab values not submitted for all patients
  mg/dl
    Blood Urea Nitrogen | 39.1 (21.3)
    Creatinine | 1.8 (0.8)
    Total Bilirubin: number analyzed (Participants) | 31
    Total Bilirubin | 1.8 (1.8)
    Plasma Free Hemoglobin: number analyzed (Participants) | 20
    Plasma Free Hemoglobin | 28.8 (28.9)
Hemodynamic Values [Mean (Standard Deviation); unit: mmHg] — Population: Hemodynamics were unable to be collected on all patients
  mmHg
    Systolic Blood Pressure: number analyzed (Participants) | 30
    Systolic Blood Pressure | 98.6 (23.2)
    Diastolic Blood Pressure: number analyzed (Participants) | 30
    Diastolic Blood Pressure | 54.2 (12.7)
    Pulmonary Artery Systolic: number analyzed (Participants) | 22
    Pulmonary Artery Systolic | 37.3 (14.0)
    Pulmonary Artery Diastolic: number analyzed (Participants) | 22
    Pulmonary Artery Diastolic | 22.9 (8.5)
    Central Venous Pressure: number analyzed (Participants) | 26
    Central Venous Pressure | 16.3 (8.0)
Glasgow Coma Scale [Count of Participants; unit: Participants]
  Eye Opening : Not done | 2
  Eye Opening : No response | 17
  Eye Opening : Response to speech | 3
  Eye Opening : Spontaneous eye opening | 10
  Motor response: Not done | 2
  Motor response: No response to pain | 13
  Motor response: Withdrawal to pain stimuli | 2
  Motor response: Localizes pain | 1
  Motor response: Obeys commands | 14
  Verbal response: Not done | 2
  Verbal response: No verbalization | 19
  Verbal response: Normal conversation | 11
Body Surface Area [Mean (Standard Deviation); unit: Meters squared] | 2.05 (0.25)
Cardiac Index [Mean (Standard Deviation); unit: L/min/m^2] — Population: Hemodynamics were unable to be collected on all patients
  L/min/m^2
    number analyzed (Participants) | 10
    (all) | 1.6 (0.4)
Cardiac Output [Mean (Standard Deviation); unit: L/min] — Population: Hemodynamics were unable to be collected on all patients
  L/min
    number analyzed (Participants) | 11
    (all) | 3.9 (1.3)
Respiratory Rate [Mean (Standard Deviation); unit: Breaths per minute] — Population: Respiratory rate data not submitted for two patients
  Breaths per minute
    number analyzed (Participants) | 30
    (all) | 17.6 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Number of patients alive 30 days after device implantation
Time Frame: 30 days post-support or to hospital discharge, whichever is longer OR to induction of anesthesia for implantation of a long-term device or heart transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Supported by the CentriMag Ventricular Assist System
Number analyzed (Participants) | 32
Participants | 20

2. Secondary Outcome: Improvement in Central Venous Pressure (CVP) and Mean Arterial Blood Pressure (MAP)
Description: Change in mean CVP while on pump support and in MAP during pump support. CVP and MAP were measured daily during pump support and the mean CVP and MAP during pump support were compared to baseline. Mean CVP or MAP during support (up to 30 days) minus baseline CVP or MAP.
Time Frame: Mean CVP or MAP during support (up to 30 days) minus baseline CVP or MAP
Population: measurements not made in all subjects
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects Supported With CentriMag
Number analyzed (Participants) | 32
mmHg
  CVP: number analyzed (Participants) | 5
  CVP | -5.5 (4.1)
  Mean arterial pressure | 7.7 (11.9)

ADVERSE EVENTS:
Time Frame: From CentriMag implant, during support, and for 6 months post device-removal
Arm/Group | Patients Supported by the CentriMag Ventricular Assist System
All-Cause Mortality (participants affected / at risk) | 15/32
Serious Adverse Events (participants affected / at risk) | 32/32
Other Adverse Events (participants affected / at risk) | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Supported by the CentriMag Ventricular Assist System (N=32)
Major bleeding (Blood and lymphatic system disorders) | 26 (73)
Cardiac arrhythmias (Cardiac disorders) | 11 (13)
Pericardial fluid collection (Cardiac disorders) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 4 (4)
Hepatic dysfunction (Hepatobiliary disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Major infection (Infections and infestations) | 13 (22)
Myocardial infarction (Cardiac disorders) | 0 (0)
Neurologic dysfunction (Nervous system disorders) | 0 (0)
Psychiatric episode (Psychiatric disorders) | 2 (2)
Renal dysfunction (Renal and urinary disorders) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Right heart failure (Cardiac disorders) | 2 (2)
Arterial non-CNS thromboembolism (Vascular disorders) | 1 (1)
Venous thromboembolism (Blood and lymphatic system disorders) | 1 (1)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1)
Other adverse event (General disorders) | 6 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Supported by the CentriMag Ventricular Assist System (N=32)
Other adverse events (General disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No